CLINICAL TRIAL: NCT04437966
Title: Assessing Effectiveness of a Chronic Disease Self-management Program in Faith-based Organizations in Barbados: a Cluster Randomized Trial
Brief Title: Chronic Disease Self-management Program for Hypertension Control in Churches
Acronym: CHIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Natasha Sobers, Lecturer, Epidemiology, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLSCHP-2008
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Twelve faith based organizations will be chosen from an organization known as New Testament Church of God Assemblies (a Pentecostal religion). Of the 12 organizations selected to participate in the study, six will be randomized to receive the intervention and six will receive usual care. the study statistician will randomly assign each church to either intervention or control groups based on a 1:1 ratio, using a pre-specified random number generator (Stata statistical software version 16). Using a 3-church block, we will assign 2 churches to intervention and 2 churches to control in each randomization block. Block randomization will be used to ensure balanced distribution of intervention and control churches.
Masking Description: Data collectors will be blinded to church randomization status until the end of the six-week recruitment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management Group (Experimental): The intervention consists of three levels - (1) chronic disease self-management workshops, (2) distribution of and teaching on the use of medication pill boxes and (3) use of social media (WhatsApp version 2.0) to encourage medication adherence.
  We combine the Stanford Chronic Disease Self-Management Curriculum, add medication adherence tools and social media use to develop a novel intervention aimed at better blood pressure control. The CDSMP focuses on enhancing skills through problem solving and brainstorming activities. In the workshop we discuss: blood pressure control, finding and affording healthy foods, label reading, physical activity, planning a healthy plate, making traditional foods healthy and portion control. Pill boxes will be distributed to all individuals in the intervention group. Post workshop, participants will be sent twice weekly reminders to use their high blood pressure medications via the social media tool WhatsApp. These will be sent for one month.
  Interventions: Behavioral: Enhanced Chronic Disease Self-management program
- Usual care group (No Intervention): Controls will receive educational material at baseline and one didactic session (on importance of medication adherence to hypertension control) lasting 1 hour delivered by a health care professional.

INTERVENTIONS:
Behavioral: Enhanced Chronic Disease Self-management program — CDSMP workshops will last for approximately 2.5 hours and occur weekly for six weeks. Sessions will focus on appropriate diet for persons with hypertension and to facilitate weight loss; managing medications, adherence to medical clinic appointments; physical activity and stress management. Participants make weekly action plans, share experiences, and help each other solve problems they encounter in creating and carrying out their self-management program. Participants will also be given pill boxes and will be prompted by social media messages to make and keep clinic appointments as well as maintain a healthy lifestyle.
  Arms: Self-management Group

SUMMARY:
In Barbados, levels of hypertension are high (40.7%) and cause of a high proportion of deaths due to cardiovascular diseases. In this study, the Stanford University-led Chronic Disease Self-Management Program (CDSMP) will be modified to form one of the basic components of a three-pronged intervention to improve blood pressure control.

Our overall goal is to evaluate the effectiveness of a hypertension self-management program in community-based settings. With the advent of the Coronavirus disease 2019 (COVID-19) we recognize that it may be necessary to adapt the programme to accommodate virtual delivery.

Our specific aims are to:

1. Adapt the Stanford (CDSMP) to ensure cultural appropriateness to Barbados. In view of the need to adhere to physical distance guidelines in the era of COVID-19 disease, modifications will be made to enhance virtual delivery while maintaining programme fidelity. We will engage stakeholders in performing modifications related to content, context and mode of delivery of the CDSMP program with the goal of ensuring cultural appropriateness.
2. Determine the clinical effectiveness of CDSMP combined with medication enhancement tools. We will conduct a cluster randomized trial in twelve faith-based organizations(FBOs) in Barbados. We are primarily interested in studying the changes in systolic blood pressure. Secondarily, we will also assess change in weight, medication adherence, dietary behavior and physical activity.
3. Understand the barriers and facilitators to implementation and sustainability of CDSMP plus self-monitoring tools in faith-based organizations. We will assess cost and sustainability of the intervention and qualitatively assess factors associated with barriers and facilitators of implementation in FBOs in Barbados.

Impact and novelty: We aim to increase the proportion of patients with controlled hypertension leading to reduced illness and deaths from strokes and heart attacks in particular. Few studies have looked at a blended approach to CDSMP delivery and these will become more necessary in the era of COVID-19. Findings on the factors impacting implementation will be transferable to small island developing states and other predominantly black populations.

DETAILED DESCRIPTION:
Setting: This cluster randomized trial will be conducted among members of selected church groups in Barbados - a small island developing state in the Caribbean with a population of approximately 287 025 (52% female). According to the Barbados' 2010 census, approximately three-quarters of the population identify as Christian. This study is intended for Christian churches in Barbados, from any denomination. Barbados is divided into 11 parishes. Given the small sizes of many churches in Barbados we have chosen to cluster by parish and divide the most densely populated parish (St. Michael) into two divisions. This gives us a total of 12 geographic divisions. Each division consists of 7-9 of our target churches comprising a total of about 350 members per division. The study will consider each division as a single unit which will be randomized to either intervention or control. The treatment of a division as one assembly allows the study to have sufficient participants at each recruitment event to be able to meet the required sample size of persons with uncontrolled hypertension.

Recruitment: Potential participants will be invited to recruitment days where they are screened for hypertension. All persons with a previous diagnosis of hypertension or currently on anti-hypertensives AND the occurrence of two or more blood pressure readings above 140 mmHg (systolic) or 90mmHg (diastolic) on the day of recruitment will be deemed eligible. Persons not known to have hypertension but who have two or more blood pressure readings above 140 mmHg (systolic) or 90mmHg (diastolic) on the day of recruitment are also eligible.

Clinical screening will also be conducted and persons will be included in the study if their systolic blood pressure (SBP) and diastolic blood pressure (DBP) readings are greater than or equal to 140 mmHg or 90 mmHg respectively on two or more readings taken at rest more than 5 minutes apart on the day of screening. Persons who are well controlled on blood pressure lowering drugs will be excluded. To obtain eligible participants, fliers and information on the study will be circulated on social media and via telephone. Recruitment days will be conducted with strict physical distancing protocols in place which are in keeping with the stage of restriction Barbados is experiencing at the time of recruitment. Recruitment will not occur during times of day time curfew and will conform to government directives.

Randomization of the churches will occur after completion of all baseline assessments, and the study statistician will randomly assign each church to either intervention or control groups based on a 1:1 ratio, using a pre-specified random number generator (Stata statistical software version 16). Using a 3-church block, we will assign 2 churches to intervention and 2 churches to control in each randomization block. Given the nature of the intervention, the trial will not be blinded. However, data collectors will be blinded to church randomization status until the end of the six-week recruitment period.

Sample size: Previous studies have found group mean SBP reductions ranging from 4.5 mmHg to 6.6 mm Hg17. Using the lowest group mean SBP reduction of 4.5 mmHg (SD 10)21 among the persons living with uncontrolled hypertension and given a study of 12 clusters we estimated that 168 persons in the intervention and 168 in the control group, would provide 80% power to detect a difference of 4.5 mmHg. This is assuming an intra-class correlation (ICC) of 0.0517. This required sample size of 336 provides us cluster sizes of 28. Given that CDSMP groups are typically between 12-16 each, we will recruit 32 per cluster (church) for a total of 192 persons in intervention and control arms each and a total required sample size of 384. Calculations were performed using Stata statistical software version 15.

Data collection (Described by aim) Aim 1: Adapt the Stanford CDSMP to ensure cultural appropriateness to Barbados: A series of stakeholder engagement meetings will be held to adapt the original lifestyle workshop series, Stanford CDSMP, so as to ensure it is culturally relevant, appropriate, and sensitive to Caribbean and Caribbean-descent populations. The Stirman et al model will be used to guide the adaptation process, allowing us to systematically look at content, context, and training adaptations. Modifications will be made to place an emphasis on medication adherence, hypertension self-management and use of the Dietary Approaches to Stop Hypertension (DASH) diet given our focus on hypertension. Foods and packaging commonly used in Barbados as well as the Caribbean Food and Nutrition Pyramids will be highlighted in the nutrition aspect of the program.

Stakeholder engagement will include researchers, dieticians, clinicians and lay persons from Barbados as well as CDSMP experts to ensure that fidelity to the essential components of the program is maintained.

Aim 2: Determine the clinical effectiveness of CDSMP combined with medication adherence tools: The intervention consists of three levels - (1) chronic disease self-management workshops, (2) distribution of and teaching on the use of medication pill boxes and (3) use of social media (WhatsApp version 2.0) to encourage medication adherence. We combine previously tested CDSMP and add medication adherence tools and social media use to develop a novel intervention focusing on improving patient self-efficacy to manage and make decisions about their illness. The Stanford-based CDSMP minimizes traditional methods of didactic knowledge transfer and focuses on enhancing skills through problem solving and brainstorming activities. In the workshop series the following will be discussed: blood pressure control, finding and affording healthy foods, label reading, physical activity, planning a healthy plate, making traditional foods healthy and portion control. These workshops are based on the Stanford Chronic Disease Self-Management Curriculum thus researchers will be trained as workshop leaders. Controls will receive educational material at baseline and one didactic session (on importance of medication adherence to hypertension control) lasting 1 hour delivered by a health care professional. Medication adherence: Pill boxes will be distributed to all individuals in the intervention group. Post workshop, participants will be sent twice weekly reminders to use their high blood pressure medications via the social media tool WhatsApp. These will be sent for a period of one month. Assessment of adherence to the patient's baseline medication before randomisation will be done by measurement of home systolic blood pressure 6 h after directly observed therapy and by returned tablet counts. Blood pressure measurements only, will be repeated after the medication adherence segment.

During an interview at the FBO, data will be collected in the following domains: demographic information (age, sex, ethnicity, education, income, address, telephone number); medication use; primary and tertiary care visit frequency; behavioral risk factors (tobacco smoking, alcohol consumption, physical inactivity, diet), medical history, place of treatment and costs incurred. Anthropometric measurements and blood pressure will be completed. Global Physical Activity questionnaire will be used as well as a food frequency questionnaire which has already been modified for use in Barbados. Questionnaires will also be used to assess self-efficacy. Immediately after the final workshop of the intervention, blood pressure, weight, physical activity survey and food frequency survey assessments will be repeated. Each control site will receive repeat measurements after the workshops are complete at the geographically closest intervention site. At each intervention site and control site, patients will be contacted six months after the first day of their workshop for repeat of weight, blood pressure, dietary habits, physical activity, medication adherence and self-efficacy. The mode of survey interviews will be face-to-face ideally. Participants will be given an electronic device and assisted with completing the survey if necessary. Participants will be given appointments to ensure that directives regarding the number of persons in the room can be adhered to. This will decrease the contact with data collectors/supporters. If however, directives from the government prevent face-to-face interviews, surveys will be done virtually.

Workshops may have to be modified to be either partially or completely online to accommodate physical distancing measures required by COVID-19 directives in place at the time of the study.

Distribution of pill boxes Each participant will be given a pill box and taught how to use these The combination of medication adherence reminders, tool box distribution and CDSMP is novel Medication adherence reminders (mHealth) Planned use of an open source, web-based social media platform (eg. WhatsApp) Others have used one-way tools like Short Message Service (SMS) texting and custom-built apps. This method will allow a secondary assessment of the impact of social interaction facilitated by WhatsApp

Aim 3: Understand the barriers and facilitators to implementation and sustainability of CDSMP plus medication adherence tools in faith-based organizations: We will focus on evaluating the implementation process by measuring fidelity, costs and sustainability. CDSMP trained master trainers will attend at least two workshops in each series to measure the extent to which workshop leaders successfully carried out the workshops as designed in Aim 1. We will track the actual cost of workshop implementation including tools needed for delivery. We will use the Program Sustainability Assessment Tool developed by the Center for Population Health Sciences, Washington University(Appendix 4) and used by the Center for Disease Control and Prevention. Leaders of the FBOs or their designate will undergo a virtual interview where this tool will be used. Interviews will be audio recorded.

Data management, safety and confidentiality: All quantitative data will be collected using Computer-Assisted Personal Interviews (CAPI), directly onto a tablet computer. The data collection infrastructure will use REDCap (a secure web application for building and managing online surveys and databases). While REDCap can be used to collect virtually any type of data, it is specifically geared to support online and offline data capture for research studies and operations. Quantitative data will be de-identified before being cleared for analysis and analyzed data will be aggregated at all times. Data analysis: We will determine the mean changes in SBP levels (primary endpoint) for the intervention group versus the control and compare differences in outcomes using mixed effects regression models. This model will allow for the effect of clustering on the precision of the estimates while allowing also for adjustment of covariates. We will adopt the intention-to-treat principle to analyze the data collected. Secondary outcomes will be assessed as follows: mean change in weight (kg) will be compared between intervention and control groups after adjustment for covariates. Changes in dietary behavior will be monitored by the calculation of the DASH diet score. Physical activity will be measured by comparing the intervention group median physical activity in MET-minutes per week. Self-efficacy scores will be calculated. Both primary and secondary outcome measures will be performed pre-implementation, immediately post-workshop and 6 months post-workshop. Quantitative assessment of fidelity and sustainability assessments will be completed calculating proportion of organizations/workshops which adhere to items on each tool. The semi-structured interviews conducted for aim 3 will be audio recorded, transcribed verbatim and analyzed using thematic content analysis to allow themes on facilitators and barriers of implementation to emerge.

ELIGIBILITY:
Inclusion Criteria:

* Resident in Barbados for the previous six months
* No plans to migrate over the ensuing one year.
* All persons with a previous diagnosis of hypertension or currently on anti- hypertensives AND the occurrence of two or more blood pressure readings above 140 mmHg (systolic) or 90mmHg (diastolic) on the day of recruitment will be deemed eligible.
* Persons not known to have hypertension but who have two or more blood pressure readings above 140 mmHg (systolic) or 90mmHg (diastolic) on the day of recruitment are also eligible

Exclusion Criteria:

* Non-residents of Barbados
* Persons whose systolic blood pressure is below 140mmHg AND/OR diastolic blood pressure below 90mmHg
* Persons who are pregnant of planning to become pregnant over the following nine months
* Unwillingness/inability to comply with the study protocol
* Current participation in another study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Six months
  We will measure systolic blood pressure before and 6 months after the interventions

SECONDARY OUTCOMES:
Mean weight change for intervention and control groups | Six months
  We will measure participants' weight in kilograms before and six months after the intervention
Level of adherence to the Dietary Approaches to Stop Hypertension (DASH) Diet | Six months
  Changes in dietary behavior will be monitored by using the Dietary Approaches to Stop Hypertension Accordance Score. Score ranges from 0 to 9. A low score represents a poor diet for hypertension control. The higher the score the more appropriate for hypertension control.
Assessing physical activity levels using the Global Physical Activity Questionnaire (GPAQ) | Six months
  Using the results of the Global Physical Activity Questionnaire median physical activity in MET-minutes per week will be calculated before the intervention as well as six months post intervention
Self-Efficacy for Managing Chronic Diseases 6-item Scale | Six months
  Perceived self-efficacy scores will be calculated using a tool developed by K Lorig(Stanford University School of Medicine) for measuring self-efficacy in chronic disease management programs. Score ranges from 1 to 10. A higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha P Sobers, PhD, Principal Investigator — George Alleyne Chronic Disease Research Centre; Lisa Brathwaite-Graham, MPH, Study Director — George Alleyne Chronic Disease Research Centre
Locations (1):
- George Alleyne Chronic Disease Research Centre, Bridgetown, Barbados

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, with standard removal of identifiable information (list the variables) and with de-identification of all dates by random shifting.
  All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available two years after the study analysis is complete.
Access Criteria: IPD will only be shared if the absolute number of participants is greater than 20. There will be grouping of variables (such as exact age) that may contribute to "potential identifiability" of participants. Researchers will be given the option of contact with PI to use original dataset for approved research purposes.

REFERENCES:
- [Derived] Sobers NP, Hambleton IR, Hassan S, Anderson SG, Brathwaite-Graham L, Lewis K, Ferguson TS. Assessing the effectiveness and implementation of a chronic disease self-management programme in faith-based organisations in Barbados: protocol for a cluster randomised parallel trial. BMJ Open. 2021 Oct 4;11(10):e050548. doi: 10.1136/bmjopen-2021-050548. PMID 34607863